CLINICAL TRIAL: NCT03307395
Title: Middle Meningeal Artery Embolization for Treatment of Chronic Subdural Hematoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1611017746
Record Dates: First submitted 2017-09-28; First posted 2017-10-11 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2020-02

CONDITIONS: Chronic Subdural Hematoma
Keywords: Chronic Subdural Hematoma; Embolization; Middle meningeal artery
MeSH Terms: conditions — Hematoma, Subdural, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Middle Meningeal Artery Embolization (Experimental)
  Interventions: Procedure: Middel Meningeal Artery Embolization

INTERVENTIONS:
Procedure: Middel Meningeal Artery Embolization — Blood supply to the subdural hematoma via the middle meningeal artery is interrupted.
  Other Names: MMA

SUMMARY:
Middle meningeal artery (MMA) embolization via a minimally invasive endovascular approach has been attempted with the goal of eliminating the arterial supply to the vascularized membrane. The investigators have recently presented the first known case series of MMA embolization as upfront treatment for cSDH in lieu of surgical evacuation (publication pending). Five patients underwent successful embolization of the MMA with subsequent reduction in size or complete resolution of cSDH with no peri-procedural complications.

The purpose of this study will be to evaluate the safety and efficacy of MMA embolization compared to traditional surgical management for symptomatic, chronic, and medically refractory SDH. MMA embolization is an established procedure used routinely for treatment of tumors or vascular malformations; this study investigates the use of an established procedure for a new disease. The investigators hypothesize that MMA embolization will afford a particularly fragile patient population an alternative to invasive and morbid neurosurgical intervention.

DETAILED DESCRIPTION:
The purpose of this study will be to evaluate the safety and efficacy of middle meningeal artery (MMA) embolization compared to traditional surgical management for symptomatic, chronic, and medically refractory subdural hematoma (SDH). MMA embolization is an established procedure used routinely for treatment of tumors or vascular malformations; this study investigates the use of an established procedure for a new disease. The investigators hypothesize that MMA embolization will afford a particularly fragile patient population an alternative to invasive and morbid neurosurgical intervention.

Since subjects being enrolled will be those that are symptomatic from chronic SDH, pre-procedural data such as clinical history, neurologic examination, and CT scans will already be available. The day after the embolization, subjects will undergo a clinical interview to assess change in symptoms. A neurologic exam and CT scan will also be performed prior to discharge. Telephone surveys will be used at intermittent time points to assess for change in clinical symptoms. The subjects will also present in clinic for a follow up clinical interview, neurologic exam, and CT scan at 2 and 6 weeks post-procedure. This follow up care including the CT scans is considered standard of care for patients undergoing surgery for chronic SDH and it will not expose them to any additional tests or imaging studies.

MMA embolization is done under moderate sedation or general anesthesia using biplane fluoroscopy. Briefly, common femoral artery access is obtained, and a guide catheter is advanced into the external carotid artery. A microcatheter is then advanced into the internal maxillary artery and then the MMA. Particles are then injected. A post-procedure carotid angiography is performed to ensure no reflux of particles into the internal carotid artery circulation. The guide catheter is then removed and femoral hemostasis is obtained. Subjects recover from anesthesia and are observed overnight, undergo a non-contrast head CT the next day, and discharged if appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Age must be greater or equal to 18 years of age.
* Subjects must have a diagnosis of chronic or acute-on-chronic subdural hematoma based on brain imaging, as documented by an independent radiologist.
* One or more symptoms attributable to chronic SDH including headache, cognitive impairment, gait instability, seizure, or mild focal neurologic deficit.
* In the opinion of the site investigator or the subject's referring physician, the subject has failed conservative management.

Exclusion Criteria:

* The subdural hematoma is causing mass effect significant enough to cause marked or progressive neurologic impairment.
* Any requirement for urgent surgical evacuation is necessary.
* Life expectancy is less than 6 months in the opinion of the subject's primary physician.
* Markedly tortuous vasculature precluding safe endovascular access, as assessed on angiogram.
* Acute subdural hematomas.
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Changes in neurological status after embolization of the MMA for symptomatic, chronic, and medically refractory SDH. | The neurological exam will be performed before the procedure, the day after the procedure, and at 2 and 6 weeks post-procedure to assess any changes in neurological status.
  A neurological exam will be performed to assess any neurological changes post-procedure.
Changes in size of the SDH post-procedure. | A head CT will be performed to assess the size of the SDH post-procedure. This will occur before the procedure, the day after the procedure, and at 2 and 6 weeks post-procedure.
  A CT scan will be performed to assess the size of the SDH before and after the procedure.

SECONDARY OUTCOMES:
The safety of embolization of the MMA for symptomatic, chronic, and medically refractory SDH | Pre-procedure, 1 day post-procedure, and 2 and 6 weeks post-procedure.
  A neurologic exam will be performed to assess any neurological deficits and/or improvements post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Jared Knopman, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data for primary and secondary outcome measures will be available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available within one year of study completion
Access Criteria: Data access requests will be reviewed by the PI.